CLINICAL TRIAL: NCT03051152
Title: Limited Versus Extended Lymphadenectomy in High Risk Elderly With Gastric Adenocarcinoma: a Randomized Controlled Trial
Brief Title: D1 Versus D2 Lymphadenectomy in High Risk Elderly With Gastric Adenocarcinoma
Acronym: LELEGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Italian Research Group for Gastric Cancer (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Varese3
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Gastric Cancer; Locally Advanced Malignant Neoplasm; Perioperative/Postoperative Complications
MeSH Terms: conditions — Stomach Neoplasms; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elderly with CCS>5 - D1 gastrectomy (Experimental): Patients aged >75 years with Charlson Comorbidity Score > 5 undergoing gastrectomy with limited lymphadenectomy
  Interventions: Procedure: D1 gastrectomy
- Elderly with CCS>5 - D2 gastrectomy (Experimental): Patients aged >75 years with Charlson Comorbidity Score > 5 undergoing gastrectomy with extended lymphadenectomy
  Interventions: Procedure: D2 gastrectomy

INTERVENTIONS:
Procedure: D1 gastrectomy — Gastrectomy with limited lymph node dissection
  Arms: Elderly with CCS>5 - D1 gastrectomy
Procedure: D2 gastrectomy — Gastrectomy with extended lymph node dissection
  Arms: Elderly with CCS>5 - D2 gastrectomy

SUMMARY:
Background: Literature often shows limited and discordant data regarding the prognostic value of age in gastric-cancer patients. Generally, disease-specific survival does not seem to be worse in the elderly when compared with younger patients, and therefore gastrectomy with extended lymphadenectomy for non-early tumors is considered the "standard" surgical therapy for all of operable patients, despite any age- or comorbidity-related limitations. Recent trials reported a survival benefit for extended nodal dissection compared with the more limited method, but some Authors found age (and comorbidities) to be a relevant predictor of postoperative complications, conditioning the safety of the surgical procedure itself.

Methods/Design: The LELEGA Trial (Limited versus Extended Lymphadenectomy in high risk Elderly with Gastric Adenocarcinoma) is a randomized, clinical multicenter trial. All patients >75 years and with Charlson Comorbidity Score >5 with resectable M0 gastric cancer are eligible for inclusion and randomization. The primary endpoint is 5-year Disease-Specific Survival (DSS). Secondary endpoints include 5-year Overall Survival (OS) and postoperative complications classified according to Clavien-Dindo. Assuming an alpha (two-sided) of 5%, 232 patients per group are necessary to achieve an 80% power to detect a 13% survival difference (from 56% to 69%) between groups.

Discussion: LELEGA trial is a prospective, multicenter randomized study to define optimal extent of lymphadenectomy (extended versus limited) in elderly and high-comorbidity gastric cancer patients.

DETAILED DESCRIPTION:
Background Although worldwide incidence of gastric cancer has decreased, it still remains the fourth most common type of cancer and the second leading cause of cancer-related death, with a growing prevalence in the elderly owing to increased life expectancy. The Literature often shows limited and discordant data regarding the prognostic value of age in gastric-cancer patients. Generally, disease-specific survival does not seem to be worse in the elderly when compared with younger patients. This evidence leads to the standardization of surgery in gastric cancer patients, whatever the age (and comorbidity). Gastrectomy with extended lymphadenectomy for non-early tumors is considered the "standard" surgical therapy for operable patients, despite any age- or comorbidity-related limitations. Following the initial doubts concerning its safety in the first randomized controlled studies, extended lymphadenectomy in gastric-cancer surgery now shows good results. Recent trials, minimizing the impact of nodal dissection on early postoperative outcome, showed a survival benefit for extended nodal dissection compared with the more limited method, particularly in advanced stages. Some of these studies showed age (and comorbidities) to be a relevant predictor of postoperative complications, conditioning the safety of the surgical procedure itself.

In a retrospective multicenter study, we examined 1.322 non-metastatic gastric-cancer patients that underwent curative gastrectomy with D2 versus D1 lymphadenectomy from January 2000 to December 2009. Postoperative complications, overall survival (OS), and disease-specific survival (DSS) according to age and the Charlson Comorbidity Score (CCS) were analyzed in relation to the extent of lymphadenectomy.

Postoperative morbidity was 30.4%. Complications were more frequent in high-morbidity elderly patients, and, although general morbidity rates after D2 and D1 lymphadenectomy were similar (29.9% and 33.2%, respectively), they also increased following D2 in high-morbidity elderly patients (39.6%). D2-lymphadenectomy significantly improved 5-year OS and DSS (48.0% vs. 37.6% in D1, p<0.001 and 72.6% vs. 58.1% in D1, p<0.001, respectively) in all patients. In elderly patients, this benefit was present only in 5-year DSS. D2 nodal dissection induced better 5-year OS and DSS rates in elderly patients with positive nodes (29.7% vs. 21.2% in D1, p=0.008 and 47.5% vs. 30.6% in D1, p=0.001, respectively), although it was present only in DSS when high-morbidity elderly patients were considered.

Even if promising, these results are derived by a retrospective study with some unavoidable biases: particularly, the selection bias depending on the choice of surgeons to perform a D1 in most elderly considered in the analysis (23.8% vs 14.4% of D1 in younger patients, p<0.001) and the unmeasurable effect of the adjuvant treatments.

Hence, a phase-III randomized controlled trial could be useful to obtain reliable data about relevant topic.

Rationale With the aging of world population, in next years we will have to face with a greater number of elderly patients. Actually, also concerning gastric cancer, this part of population is usually excluded from clinical trial, and hence guidelines are not "tested" for them. Many retrospective studies (including our retrospective analysis on a very large series) did not solve any doubt about short-term outcomes and survival benefit of D2 gastrectomy in high-risk elderly patients. Evident methodological limitations limit the relevance of their conclusions. Firstly, the retrospective design of these studies implies non-homogeneous groups, unavoidably influenced by the different cut-offs used for "elderly" definition and by the surgeons' choice with particular regard to lymphadenectomy. Secondly, they often did not consider any adjuvant therapy: although analysis would have been influenced by the administration of different regimens with different schedules, survival might have been modified, thus conditioning the interpretation of results. According the results of these retrospective reports extended lymphadenectomy confirmed its efficacy in determining better survival rates in gastric cancer patients. However, after extended nodal dissection OS in high-morbidity elderly patients, even with nodal involvement, does not present undoubted benefits. Most of these studies did not have sufficient power to validate their conclusions.

In conclusion, this prospective randomized multicenter trial will test the effect of extension of lymphadenectomy on the particular setting of high-risk elderly patients in the attempt to identify those patients most likely to benefit from aggressive radical surgery with acceptable perioperative risk.

STUDY DESIGN This is a multicenter, open randomized trial

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >75 years, with CCS >5, undergoing curative surgery for locally advanced M0 gastric adenocarcinoma. All patients aged >75 years with a Charlson Comorbidity Score (CCS) [17] of at least 5, with an endoscopic and histological diagnosis of gastric adenocarcinoma underwent standard preoperative staging: contrast enhanced computed tomography of chest, abdomen (with gastric distention) and pelvis. Preoperative staging laparoscopy should be performed in order to exclude peritoneal carcinomatosis.
* Patients with ability to understand the nature or consequences of the trial.
* Patients with ability to provide written informed consent.

Exclusion Criteria:

* Previous surgery of the stomach.
* Patients with a previous history of cancer (< 5 year) or presenting with a co-existing cancer.
* Patients with bulky nodes at the second level stations;
* Patients requiring multi-organ resection;
* Patients refusing blood transfusions;
* Patients recruited for other trial;
* Patients operated in an acute setting are excluded to allow for appropriate inclusion and randomization.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
5y-DSS | 5 years
  5-year Disease-Specific Survival (DSS)

SECONDARY OUTCOMES:
5y-OS | 5 years
  5-year Overall Survival (OS)
Post-operative complications | 30 days
  Post-operative complications according to Clavien Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Rausei, MD, PhD, Principal Investigator — ASST Settelaghi - University of Insubria
Locations (1):
- ASST Settelaghi - University of Insubria, Varese, Varese, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Rausei S, Ruspi L, Rosa F, Morgagni P, Marrelli D, Cossu A, Cananzi FC, Lomonaco R, Coniglio A, Biondi A, Cipollari C, Graziosi L, Fumagalli U, Casella F, Bertoli P, di Leo A, Alfieri S, Vittimberga G, Roviello F, Orsenigo E, Quagliuolo V, Montemurro S, Baiocchi G, Persiani R, Bencivenga M, Donini A, Rosati R, Sansonetti A, Ansaloni L, Zanoni A, Galli F, Dionigi G; Italian Research Group for Gastric Cancer (IRGGC). Extended lymphadenectomy in elderly and/or highly co-morbid gastric cancer patients: A retrospective multicenter study. Eur J Surg Oncol. 2016 Dec;42(12):1881-1889. doi: 10.1016/j.ejso.2016.05.003. Epub 2016 Jun 1. PMID 27266816
- [Background] Wu CW, Hsiung CA, Lo SS, Hsieh MC, Chen JH, Li AF, Lui WY, Whang-Peng J. Nodal dissection for patients with gastric cancer: a randomised controlled trial. Lancet Oncol. 2006 Apr;7(4):309-15. doi: 10.1016/S1470-2045(06)70623-4. PMID 16574546
- [Background] Degiuli M, Sasako M, Ponti A, Vendrame A, Tomatis M, Mazza C, Borasi A, Capussotti L, Fronda G, Morino M; Italian Gastric Cancer Study Group. Randomized clinical trial comparing survival after D1 or D2 gastrectomy for gastric cancer. Br J Surg. 2014 Jan;101(2):23-31. doi: 10.1002/bjs.9345. PMID 24375296
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912